CLINICAL TRIAL: NCT03068754
Title: A Multicenter, Double Blind, Placebo Controlled Study to Assess the Efficacy and Safety of H.P. Acthar® Gel in the Treatment of Subjects With Amyotrophic Lateral Sclerosis
Brief Title: Study of Acthar® Gel (Acthar) for Amyotrophic Lateral Sclerosis (ALS)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: As recommended by the study's independent Data and Safety Monitoring Board (DSMB)
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MNK14042068
Record Dates: First submitted 2017-02-23; First posted 2017-03-03 (Actual); Results first posted 2020-09-03 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to treatment group randomly (like flipping a coin). They will have a 2 out of 3 chance of receiving the study drug, and a 1 out of 3 chance of receiving placebo during the treatment period. All participants who continue into the extension period receive Acthar.
Who Masked: Participant, Investigator
Masking Description: The Treatment Period is defined as Randomized (2:1, Arm A: Arm B), Double-blind (with care provider and outcomes assessor also blinded).
  The Extension Period has no masking, because all who participate receive open label study drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: Treatment Period Acthar (Experimental): Participants receive one 0.2 mL subcutaneous (SC) injection (shot under the skin) of the study drug (Acthar), daily for up to 36 weeks.
  Those who do not continue into the extension period will have 3 weeks of tapering off the drug, ending their participation by Week 39.
  Interventions: Drug: Acthar
- Arm B: Treatment Period Placebo (Placebo Comparator): Participants receive one 0.2 mL SC injection that looks like Acthar, but has no drug in it (Matching Placebo), daily for up to 36 weeks.
  Those who do not continue into the extension period will have 3 weeks of simulated tapering, ending their participation by Week 39.
  Interventions: Drug: Placebo
- Arm C: Extension Period Acthar-Acthar (Experimental): Participants who receive Acthar during the treatment period and continue into the extension period do not go through the treatment-period tapering, but receive one 0.2 mL SC injection of Acthar, daily for up to 48 weeks, followed by 3 weeks of tapering off the drug, ending their participation within about 21 months.
  Interventions: Drug: Acthar
- Arm D: Extension Period Placebo-Acthar (Experimental): Participants who receive Placebo during the treatment period and continue into the extension period do not go through the treatment-period simulated tapering, but receive one 0.2 mL SC injection of Acthar, daily for up to 48 weeks, followed by 3 weeks of tapering off the drug, ending their participation within about 21 months.
  Interventions: Drug: Acthar; Drug: Placebo

INTERVENTIONS:
Drug: Acthar — Repository corticotropin for subcutaneous injection
  Other Names: Trade name: Acthar® Gel; Generic name: repository corticotropin injection
  Arms: Arm A: Treatment Period Acthar; Arm C: Extension Period Acthar-Acthar; Arm D: Extension Period Placebo-Acthar
Drug: Placebo — Matching placebo for subcutaneous injection
  Other Names: Matching Placebo; Reference Product
  Arms: Arm B: Treatment Period Placebo; Arm D: Extension Period Placebo-Acthar

SUMMARY:
About 213 people with ALS will participate in this study. There will be locations in North and South America.

During the first part, participants will be randomly assigned to a group (like by flipping a coin). Out of every 3:

* 2 will get the study drug
* 1 will get a look-alike with no drug in it (placebo)

During the second part, everyone will get the study drug.

Participation will help doctors find out if Acthar can help or slow down the symptoms of ALS better than placebo.

DETAILED DESCRIPTION:
This is a multicenter, multiple dose study to examine the effect of Acthar on functional decline in adult participants with ALS. Approximately 213 participants will be enrolled.

Following a screening period of up to 28 days, participants with ALS and symptom onset (defined as first muscle weakness or dysarthria) ≤ 2 years prior to the Screening Visit will be randomized on a 2:1 basis to receive subcutaneous (SC) Acthar 0.2 mL (16 Units [U]) daily (QD) or SC matching placebo 0.2 mL QD for 36 weeks, followed by a 3-week taper.

Participants who complete the 36 week double-blind treatment period are eligible to enter an Open Label Extension phase in which all participants will receive Acthar 0.2 mL (16 U) daily.

ELIGIBILITY:
Inclusion Criteria:

1. Is 18-75 years of age at Screening
2. Has ALS symptom onset within 2 years prior to Screening
3. Has forced vital capacity (FVC) no higher than 60% at screening
4. If taking riluzole, is on a stable dose for 4 weeks before Screening

Exclusion Criteria:

1. Has tracheostomy, diaphragm pacing, or an ongoing need for assisted ventilation of any type
2. Has used any medication within a time period not allowed per protocol
3. Has history of Type 1 or Type 2 diabetes mellitus, or any clinically significant infection
4. Used edaravone less than 1 week before Screening
5. Received any stem cell replacement therapy
6. Used steroids within a time period not allowed per protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Mallinckrodt
Locations (69):
- United States (39):
  - Neuromuscular Research Center, Phoenix, Arizona
  - Mayo Clinic - Arizona, Scottsdale, Arizona
  - University of California San Diego, La Jolla, California
  - Loma Linda University Health System, Department of Neurology, Loma Linda, California
  - Keck School of Medicine, University of Southern California, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - University of California Irvine Medical Center, Orange, California
  - California Pacific Medical Center, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - George Washington University, Washington D.C., District of Columbia
  - University of Florida - McKnight Brain Institute, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Indiana University-Neuroscience Center of Excellence/Goodman Hall, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - John Hopkins Outpatient Center, Baltimore, Maryland
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Mercy Health- Saint Mary's, Grand Rapids, Michigan
  - Neurology Associates, Lincoln, Nebraska
  - University of Nebraska Medical Center - Physicians Clinical Neurosciences Center, Omaha, Nebraska
  - Las Vegas Clinic, Las Vegas, Nevada
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Columbia Presbyterian Hospital, New York, New York
  - Providence ALS Center, Portland, Oregon
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Wesley Neurology Clinic, Cordova, Tennessee
  - Austin Neuromuscular Center, Austin, Texas
  - Texas Neurology, P.A., Dallas, Texas
  - The Methodist Hospital, Houston, Texas
  - University of Vermont Medical Center, Colchester, Vermont
  - VCU Medical Center, Richmond, Virginia
  - Swedish Neuroscience Institute, Seattle, Washington
  - Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin
- Argentina (10):
  - IADIN, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - STAT Research, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - DIABAID, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - INEBA, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Español, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Británico de Buenos Aires, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - ILAIM, Córdoba, Córdoba Province
  - Fundación Scherbovsky, Mendoza, Mendoza Province
  - Instituto de Neurología y Neurorrehabilitación del Litoral (INNeL ), Santa Fe, Santa Fe Province
- Canada (4):
  - Edmonton Kaye Clinic, Edmonton, Alberta
  - Recherche Sepmus inc, Greenfield Park, Quebec
  - Centre de recherché du Centre Hospitalier de l'Universite de Montreal (CRCHUM), Montreal, Quebec
  - Montreal Neurological Institute & Hospital, Montreal, Quebec
- Chile (3):
  - Centro de Trastornos del Movimiento (CETRAM), Santiago, Santiago Metropolitan
  - Clinica Dávila, Santiago, Santiago Metropolitan
  - Biomedica Research Group AV Salvador 149, oficina 1101, Santiago
- Centro de Investigaciones Clínicas SAS, Cali, Colombia
- Mexico (7):
  - Clinical Research Institute Saltillo S.A. de C.V., Saltillo, Coahuila
  - Hospital Universitario "Dr. José Eleuterio González", Monterrey, Nuevo León
  - SMIQ BRCR Global México, Querétaro City, Querétaro
  - Clinical Research Institute S.C., San Lucas Tepetlacalco, Tlalnepantla De Baz
  - Centro Especializado en Investigación Clínica S.C., Boca del Río, Veracruz
  - Phylasis Clinicas Research, Mexico City
  - FAICIC Clinical Researc, Veracruz
- Peru (5):
  - Hospital Nivel IV Carlos Alberto Seguin Escobedo, Arequipa
  - Hospital Nacional IV Alberto Sabogal Sologuren, Callao
  - Hospital Almenara, Lima
  - Instituto Neuro Cardiovascular de las Américas, Lima
  - Hospital Nacional Cayetano Heredia, Lima

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 207 potential participants screened, 143 were randomized to begin treatment
Groups:
- Arm A: Randomized Treatment Period (RTP) Acthar Gel: Participants receive one 0.2 mL subcutaneous (SC) injection (shot under the skin) of the study drug (Acthar Gel), daily for up to 36 weeks.
  Those who do not continue into the extension period had 3 weeks of tapering off the drug, ending their participation by Week 39.
- Arm B: RTP Placebo: Participants receive one 0.2 mL SC injection that looks like Acthar, but has no drug in it (matching Placebo), daily for up to 36 weeks.
  Those who do not continue into the extension period had 3 weeks of simulated tapering, ending their participation by Week 39.
- Arm C: Open Label Extension Period (OLE) Acthar Gel-Acthar Gel: Participants who received Acthar Gel during the treatment period and continue into the extension period do not go through the treatment-period tapering, but receive one 0.2 mL SC injection of Acthar Gel, daily for up to 48 weeks, followed by 3 weeks of tapering off the drug, ending their participation within about 21 months.
- Arm D: OLE Placebo-Acthar Gel: Participants who received Placebo during the treatment period and continue into the extension period do not go through the treatment-period simulated tapering, but receive one 0.2 mL SC injection of Acthar, daily for up to 48 weeks, followed by 3 weeks of tapering off the drug, ending their participation within about 21 months.
Period: Randomized Treatment Period (RTP)
Arm/Group | Arm A: Randomized Treatment Period (RTP) Acthar Gel | Arm B: RTP Placebo | Arm C: Open Label Extension Period (OLE) Acthar Gel-Acthar Gel | Arm D: OLE Placebo-Acthar Gel
Started | 95 | 48 | 0 (OLE Arms were not included during the RTP) | 0
Intention to Treat (ITT) Population | 95 | 48 | 0 | 0
Safety Population | 95 | 47 | 0 | 0
Modified ITT (mITT) | 93 | 46 | 0 | 0
Completed Taper (Defined as completing the End of RTP Taper Visit at about Week 39 or an early termination visit) | 58 | 28 | 0 | 0
Completed 36 Weeks of Treatment | 28 | 9 | 0 | 0
Completed RTP (Defined as completing 36 weeks of treatment, followed by Week 39 visit or entering the OLE period) | 27 | 9 | 0 | 0
Enrolled in OLE Period | 25 | 8 | 0 | 0
Completed | 28 | 9 | 0 | 0
Not Completed | 67 | 39 | 0 | 0
Not completed — Adverse Event | 1 | 3 | 0 | 0
Not completed — Death | 2 | 2 | 0 | 0
Not completed — Disease progression | 1 | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 2 | 0 | 0
Not completed — Discontinued by Physician | 1 | 0 | 0 | 0
Not completed — Subject Decision based on Compensation | 0 | 1 | 0 | 0
Not completed — Trial Terminated by Sponsor | 55 | 29 | 0 | 0
Period: Open Label Extension Period (OLE)
Arm/Group | Arm A: Randomized Treatment Period (RTP) Acthar Gel | Arm B: RTP Placebo | Arm C: Open Label Extension Period (OLE) Acthar Gel-Acthar Gel | Arm D: OLE Placebo-Acthar Gel
Started (Safety Population in the OLE - 4 participants who completed RTP were not treated in the OLE) | 0 (RTP arms were not included during the OLE period) | 0 | 25 | 8
Completed Taper (Completed End of Taper visits after Week 84 visit or being terminated early from the OLE period) | 0 | 0 | 19 | 7
Completed OLE Period (Completed Week 84 visit, End of Taper visit and follow up visit) | 0 | 0 | 3 | 2
Completed Treatment in OLE (Completed Week 84 visit) | 0 | 0 | 4 | 2
Completed (Completed treatment in OLE period) | 0 | 0 | 4 | 2
Not Completed | 0 | 0 | 21 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Disease progression | 0 | 0 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 5 | 0
Not completed — Subject Discontinued for Non-efficacy | 0 | 0 | 1 | 0
Not completed — Trial Terminated by Sponsor | 0 | 0 | 12 | 3

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Arm A: RTP Acthar Gel: Participants receive one 0.2 mL subcutaneous (SC) injection (shot under the skin) of the study drug (Acthar Gel), daily for up to 36 weeks.
  Those who do not continue into the extension period will have 3 weeks of tapering off the drug, ending their participation by Week 39.
- Arm B: RTP Placebo: Participants receive one 0.2 mL SC injection that looks like Acthar, but has no drug in it (matching Placebo), daily for up to 36 weeks.
  Those who do not continue into the extension period will have 3 weeks of simulated tapering, ending their participation by Week 39.
- Total: Total of all reporting groups
Arm/Group | Arm A: RTP Acthar Gel | Arm B: RTP Placebo | Total
Number analyzed (Participants) | 95 | 47 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (10.80) | 56.3 (10.68) | 56.0 (10.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 21 | 56
  Male | 60 | 26 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 19 | 57
  Not Hispanic or Latino | 57 | 28 | 85
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 2 | 7
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 72 | 33 | 105
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 11 | 26

OUTCOME MEASURES:

1. Primary Outcome: Treatment Period: Scores on a Scale for Telephone-administered Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R)
Description: The ALSFRS-R is a validated questionnaire-based scale used extensively as a primary outcome measure in ALS clinical trials and is considered a predictor of survival.
  ALSFRS-R is a 12-item scale that measures 4 domains relevant for ALS (gross motor, fine motor, bulbar and respiratory)
  A trained, independent rater calls each participant (or the caregiver) to administer the questionnaire. The 12 functions are rated on a scale from 0 to 4, with a highest possible (summed) score of 48. Higher scores represent better function.
Time Frame: Baseline, Week 36
Population: Safety Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: RTP Acthar Gel | Arm B: RTP Placebo
Number analyzed (Participants) | 95 | 47
score on a scale
  Baseline | 34.7 (6.01) | 34.3 (5.84)
  Week 36: number analyzed (Participants) | 27 | 9
  Week 36 | 26.4 (9.34) | 30.8 (7.55)

2. Primary Outcome: Number of Participants Experiencing an Adverse Event During the Treatment Period
Description: Serious adverse events, non-serious treatment-emergent adverse events, and all-cause mortality are collected until the participant no longer participates in the study Clinically significant changes in safety measures are recorded as adverse events.
Time Frame: by the end of the treatment period (within 36 Weeks)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: RTP Acthar Gel | Arm B: RTP Placebo
Number analyzed (Participants) | 95 | 47
Participants
  Serious Treatment Emergent Adverse Events | 13 | 6
  Non-serious Treatment-Emergent Adverse Events | 74 | 40
  Death | 2 | 3

3. Primary Outcome: Number of Participants Experiencing an Adverse Event by the End of the Trial in the OLE Period
Description: Serious adverse events, non-serious treatment-emergent adverse events, and all-cause mortality are collected until the participant no longer participates in the study (estimated about 1 year for participants leaving after the treatment period, and two years for participants who participate also in the open label extension). Clinically significant changes in safety measures are recorded as adverse events.
Time Frame: by the time of database lock (within 84 weeks)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Arm C: OLE Acthar Gel-Acthar Gel: Participants who receive Acthar Gel during the treatment period and continue into the extension period do not go through the treatment-period tapering, but receive one 0.2 mL SC injection of Acthar Gel, daily for up to 48 weeks, followed by 3 weeks of tapering off the drug, ending their participation within about 21 months.
- Arm D: OLE Placebo-Acthar Gel: Participants who receive Placebo during the treatment period and continue into the extension period do not go through the treatment-period simulated tapering, but receive one 0.2 mL SC injection of Acthar, daily for up to 48 weeks, followed by 3 weeks of tapering off the drug, ending their participation within about 21 months.
Arm/Group | Arm C: OLE Acthar Gel-Acthar Gel | Arm D: OLE Placebo-Acthar Gel
Number analyzed (Participants) | 25 | 8
Participants
  Serious Treatment Emergent Adverse Events | 4 | 2
  Non-serious Treatment-Emergent Adverse Events | 20 | 7

4. Secondary Outcome: Treatment Period: Spirometry (%)
Description: Spirometry (meaning the measuring of breath) is the most common of the lung function tests. It measures how much air can be inhaled [Forced Vital Capacity (FVC)] and exhaled [(Forced Expiratory Volume in one second (FEV1)].
Time Frame: Baseline, Week 36
Population: Safety population
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Arm A: RTP Acthar Gel | Arm B: RTP Placebo
Number analyzed (Participants) | 95 | 47
liters
  FVC at Baseline | 85.0 (18.31) | 82.1 (17.60)
  FVC at Week 36: number analyzed (Participants) | 27 | 8
  FVC at Week 36 | 61.4 (27.37) | 63.8 (26.05)
  FEV1 at Baseline | 79.3 (18.78) | 77.8 (18.52)
  FEV1 at Week 36: number analyzed (Participants) | 27 | 8
  FEV1 at Week 36 | 59.1 (27.37) | 54.3 (26.79)

5. Secondary Outcome: Treatment Period: Scores on a Scale for Investigator-administered ALSFRS-R
Description: The ALSFRS-R is a 12-item scale evaluating 4 domains relevant to ALS (gross motor, fine motor, bulbar and respiratory).
  The trained investigator (or designee) administers the ALSFRS-R questionnaire in person with the participant (or caregiver). The 12 functions are rated on a scale from 0 to 4, with a highest possible (summed) score of 48. Higher scores represent better function.
Time Frame: Baseline, Week 36
Population: Safety Population, with an actual score at the given time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: RTP Acthar Gel | Arm B: RTP Placebo
Number analyzed (Participants) | 95 | 47
score on a scale
  Baseline: number analyzed (Participants) | 93 | 45
  Baseline | 35.8 (6.05) | 35.4 (6.23)
  Week 36: number analyzed (Participants) | 29 | 9
  Week 36 | 28.0 (9.50) | 30.9 (7.18)

6. Secondary Outcome: Extension Period: Scores on a Scale for Investigator-administered ALSFRS-R
Description: The ALSFRS-R is a 12-item scale evaluating 4 domains relevant to ALS (gross motor, fine motor, bulbar and respiratory).
  The trained investigator (or designee) administers the ALSFRS-R questionnaire in person with the participant (or caregiver). The 12 functions are rated on a scale from 0 to 4, with a highest possible score of 48. Higher scores represent better function.
Time Frame: Baseline, Week 84
Population: OLE population with scores at the given week; baseline is defined as the value at randomization (week 0)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm C: OLE Acthar Gel-Acthar Gel | Arm D: OLE Placebo-Acthar Gel
Number analyzed (Participants) | 25 | 7
units on a scale
  Baseline | 36.8 (5.33) | 39.6 (1.81)
  Week 84: number analyzed (Participants) | 5 | 2
  Week 84 | 27.4 (5.41) | 21.5 (4.95)

ADVERSE EVENTS:
Time Frame: From the start to the end of the period; RTP is 36 weeks (plus 3 weeks if ending there), OLE is up to 21 months (up to Week 84)
Description: Treatment-emergent adverse events (TEAEs) were collected. A TEAE is defined as an adverse event that starts or worsens on or after first dose of study drug and within 28 days from the last dose date of the study drug (For subjects entered into OLE, any TEAE started prior to first OLE dose is counted in RTP). For each system organ class and preferred term, subjects are counted only once, even if they experienced multiple events in that system organ class or preferred term.
Arm/Group | Arm A: RTP Acthar Gel | Arm B: RTP Placebo | Arm C: OLE Acthar Gel-Acthar Gel | Arm D: OLE Placebo-Acthar Gel
All-Cause Mortality (participants affected / at risk) | 2/95 | 3/47 | 1/25 | 2/8
Serious Adverse Events (participants affected / at risk) | 13/95 | 6/47 | 4/25 | 2/8
Other Adverse Events (participants affected / at risk) | 71/95 | 34/47 | 18/25 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: RTP Acthar Gel (N=95) | Arm B: RTP Placebo (N=47) | Arm C: OLE Acthar Gel-Acthar Gel (N=25) | Arm D: OLE Placebo-Acthar Gel (N=8)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 0 (0) | 1 (1) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: RTP Acthar Gel (N=95) | Arm B: RTP Placebo (N=47) | Arm C: OLE Acthar Gel-Acthar Gel (N=25) | Arm D: OLE Placebo-Acthar Gel (N=8)
Constipation (Gastrointestinal disorders) | 13 (15) | 4 (5) | 2 (3) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 5 (5) | 0 (0) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 5 (5) | 5 (5) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (6) | 2 (2) | 2 (2) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 5 (6) | 1 (1) | 0 (0) | 1 (1)
Asthenia (General disorders) | 6 (7) | 4 (5) | 1 (1) | 1 (1)
Fatigue (General disorders) | 13 (14) | 6 (8) | 3 (3) | 1 (1)
Injection site bruising (General disorders) | 13 (16) | 4 (6) | 0 (0) | 0 (0)
Oedema (General disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 17 (24) | 2 (2) | 2 (2) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 8 (12) | 2 (2) | 4 (6) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 9 (14) | 2 (4) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 18 (28) | 14 (33) | 6 (11) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 5 (7) | 1 (1) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 3 (3) | 5 (6) | 1 (1) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (16) | 4 (8) | 0 (0) | 1 (1)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (5) | 3 (3) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 (16) | 3 (3) | 2 (3) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 22 (35) | 9 (14) | 3 (3) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 7 (7) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (4) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 7 (7) | 3 (3) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 9 (12) | 4 (5) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 11 (14) | 1 (6) | 1 (1) | 2 (2)
Muscle contractions involuntary (Nervous system disorders) | 3 (3) | 3 (3) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 6 (6) | 2 (3) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 3 (4) | 3 (3) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 6 (8) | 1 (1) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 8 (10) | 1 (1) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 7 (7) | 1 (1) | 2 (3) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased viscosity of upper respiratory secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/54/NCT03068754/Prot_SAP_000.pdf